CLINICAL TRIAL: NCT05124392
Title: Biomarker Profiling in Individuals at Risk for Prion Disease
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Broad Institute of MIT and Harvard (Other)
Responsible Party: Principal Investigator, Steven E Arnold, MD, Professor of Neurology, Massachusetts General Hospital
Other Study IDs: 2017P000214
Record Dates: First submitted 2021-10-27; First posted 2021-11-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: CJD (Creutzfeldt Jakob Disease); Prion Diseases; GSS; FFI; Familial Fatal Insomnia
MeSH Terms: conditions — Insomnia, Fatal Familial; Prion Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Blood and Cerebral Spinal Fluid for biomarker quantification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with a family history of Prion disease: Individuals with a family history of Prion disease

SUMMARY:
We are doing this research to identify biomarkers in individuals who are at-risk for familial prion disease. We hope to use these biomarkers to predict timing of disease onset in pre-symptomatic individuals and to guide the direction of future clinical trials.

DETAILED DESCRIPTION:
This study aims to measure biomarkers longitudinally in individuals at risk of developing genetic prion disease to identify clinical assays and molecular markers that: can inform our understanding of pre-clinical pathology, predict timing of disease onset in pre-symptomatic individuals, and enable development and evaluation of novel treatment efficacy in pre-symptomatic or early symptomatic individuals.

Participation in the study involves annual visits to the clinic site in Charlestown, MA. Study visits include: a medical exam, blood draws, cognitive tests and questionnaires, spinal fluid collection, and (optional) MRI.

Travel support and stipend is provided for interested individuals.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Aged 18 - 85,
2. One of the following:

   1. Known carrier of pathogenic PRNP mutation
   2. History of probable or definite prion disease in biological parent and other family members
   3. Non-carrier family members and/or unrelated previously enrolled negative control volunteers
3. Medically safe to undergo blood draw, lumbar puncture and cognitive testing,
4. Adequate visual and auditory acuity to complete cognitive testing,
5. Fluent in English,
6. At least 5 years of education,
7. Capable of providing informed consent and following study procedures,
8. No contraindications to MRI scanning as determined via the Martinos Center MRI Screening process (for PRNP mutation carriers ONLY)

Exclusion Criteria:

1. Any CNS disease other than asymptomatic or early prion disease, such as clinical stroke, brain tumor, multiple sclerosis, significant head trauma with persistent neurological or neurocognitive deficits, Alzheimer's disease, Parkinson's disease, frontotemporal lobar degeneration or other known neurodegenerative disease,
2. History of alcohol or other substance abuse or dependence within the past two years,
3. Any significant systemic illness or unstable medical condition or pregnancy that could represent safety risk or affect participation in the study,
4. Coagulopathy or anti-coagulant therapy (such as Coumadin) increasing the risk for phlebotomy or lumbar puncture resulting in PT/PTT and INR within 1.5 standard deviation over the upper normal limit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 people ages 18-85 with history of genetic prion disease and 50 non-carrier healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
CSF YKL40 | 1 year
  Levels of YKL40
CSF Tau | 1 year
  Levels of Tau
CSF Nfl | 1 year
  Levels of Nfl
CSF GFAP | 1 year
  Levels of GFAP
CSF Prion protein | 1 year
  Levels of Prion protein
CSF Prion biomarkers | 1 year
  RT-QuIC levels
Cognition | 1 year
  NIH Toolbox measures of cognition

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Arnold, MD, Principal Investigator — MGH
Locations (1):
- Alzheimer's Clinical and Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Vallabh SM, Mortberg MA, Allen SW, Kupferschmid AC, Kivisakk P, Hammerschlag BL, Bolling A, Trombetta BA, Devitte-McKee K, Ford AM, Sather LE, Duffy G, Rivera A, Gerber J, McManus AJ, Minikel EV, Arnold SE. Fluid Biomarkers in Individuals at Risk for Genetic Prion Disease up to Disease Conversion. Neurology. 2024 Jul 23;103(2):e209506. doi: 10.1212/WNL.0000000000209506. Epub 2024 Jun 19. PMID 38896810